CLINICAL TRIAL: NCT06671223
Title: Effectiveness of Infiltrations in the Treatment of Plantar Fasciopathy: A Randomized Clinical Study.
Brief Title: Effectiveness of Infiltrations in the Treatment of Plantar Fasciopathy
Acronym: INFILTRA-PLANT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, ANA MARIA RAYO PEREZ, Principal Investigator, University of Seville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TFMAGM; TFMAGM2024 (Other: Universidad de Sevilla)
Record Dates: First submitted 2024-09-26; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Plantar Fasciitis of Both Feet; Plantar Fasciopathy
Keywords: plantar fasciitis; fasciopaty; corticosteroid; PRP; hyaluronic acid; infiltrations; treatment
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Conservative Treatment; Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups:
  Intervention group: They will receive corticosteroid infiltrations under ultrasound guidance.
  Control group: They will receive conservative treatment that may include physiotherapy and recommendations for foot care, without infiltrations.
Who Masked: Investigator
Masking Description: In this study, a double-blind design is implemented to ensure data integrity and reduce bias. The following roles are masked:
  Participants: Participants are not informed to which treatment group they have been assigned (corticosteroid infiltrations or conservative treatment).
  Investigators: Investigators evaluating clinical outcomes, including pain measurement and foot function, are blinded to the treatment group assignment of participants.
  Healthcare Providers: The professionals administering the infiltrations are masked regarding treatment assignment, as a third party, not involved in the study, will be responsible for performing the infiltrations.
  Data Monitors: Data monitors monitoring the safety and integrity of the study are also blinded to treatment assignments until final analysis of the results is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corticoesteroid Infiltrations (Experimental): In this group, participants will receive infiltrations directly into the affected plantar fascia. This intervention aims to reduce the inflammation and pain associated with plantar fasciopathy.
  Interventions: Drug: Infiltration
- Conservative treatment (Placebo Comparator): Participants in this group will receive conservative treatment that does not include infiltrations. This approach is based on non-invasive methods that are commonly used to manage plantar fasciopathy.
  Interventions: Other: Conservative treatment

INTERVENTIONS:
Drug: Infiltration — The intervention consists of the administration of infiltrations in the affected plantar fascia of participants with a diagnosis of plantar fasciopathy. A drug such as a corticosteroid, PRP or hyaluronic acid will be used, which will be injected under ultrasound guidance to ensure precision at the site of the injury. This intervention aims to reduce inflammation and pain, thus improving the functionality of the foot. Up to three infiltrations will be performed, depending on the patient's response to treatment and medical evaluation. The infiltrations will be compared with a control group that will receive conservative treatment without infiltrations, to evaluate the relative effectiveness of this pharmacological intervention in the management of plantar fasciopathy.
  Other Names: Intervention group
  Arms: Corticoesteroid Infiltrations
Other: Conservative treatment — The control group is used to compare the effectiveness of infiltrations with a non-invasive approach in the treatment of plantar fasciopathy. This group will not receive any infiltration and will focus on conservative interventions.
  Other Names: Control group
  Arms: Conservative treatment

SUMMARY:
This clinical study aims to evaluate the effectiveness of infiltrations in the treatment of plantar fasciopathy, a painful condition that affects the sole of the foot and is common in active people. Plantar fasciopathy is caused by inflammation or damage to the plantar fascia, the tissue that connects the heel to the toes. Participants in this study will be randomly assigned to receive one of two treatments: corticosteroid infiltrations or conservative treatment without infiltrations. Infiltrations will be guided by ultrasound to ensure accuracy. The study will evaluate pain reduction and improvement in foot function over a six-month period. The objective of the study is to determine if infiltrations provide a significant improvement compared to other non-invasive treatments. The results will help doctors and patients make informed decisions about the best treatment options for plantar fasciopathy.

DETAILED DESCRIPTION:
This clinical study, titled "Effectiveness of Infiltrations in the Treatment of Plantar Fasciopathy", will be carried out at the University of Seville and its main objective is to evaluate the impact of corticosteroid infiltrations on pain reduction and functional improvement in patients diagnosed with plantar fasciopathy.

ELIGIBILITY:
Inclusion Criteria:

Age: Participants aged 18 to 50 years. Diagnosis: Confirmed diagnosis of plantar fasciopathy based on clinical evaluation and imaging (if applicable).

Duration of Symptoms: Symptoms persisting for at least 6 weeks prior to enrollment.

Pain Level: Reported pain level of at least 4 on the Visual Analog Scale (VAS) at baseline.

Ability to Comply: Participants must be able to follow study protocols and attend follow-up appointments.

Informed Consent: Participants must provide written informed consent to participate in the study.

Exclusion Criteria:

Other Foot Pathologies: Presence of other significant foot conditions (e.g., fractures, arthritis, tarsal tunnel syndrome) that could interfere with the study results.

Pregnancy or Breastfeeding: Pregnant or breastfeeding individuals will be excluded from the study.

Neurological Disorders: History of significant neurological disorders affecting lower limb function.

Systemic Conditions: Patients with systemic conditions (e.g., diabetes, autoimmune diseases) that could affect healing or response to treatment.

Allergy to Corticosteroids: Known allergy or adverse reaction to corticosteroids or local anesthetics.

Psychiatric Disorders: Individuals with severe psychiatric disorders that may impair their ability to provide informed consent or adhere to the study protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Level | Evaluations will be carried out at the beginning of the study, and at 3, 6 and 12 weeks after the intervention.
  Pain level will be assessed using the Visual Analogue Scale 0 to 10 points (VAS), where participants will mark their pain level on a 10 cm line, from "no pain" (0) to "unbearable pain" (10).

SECONDARY OUTCOMES:
Functional Improvement | Evaluations at the beginning, and at 3, 6 and 12 weeks post-intervention.
  Foot functionality will be assessed using the Foot Function Index 0 to 100 points (FFI), which measures the functional capacity of the foot and the impact of pain on daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: No